CLINICAL TRIAL: NCT01679223
Title: Objective Evaluation of Collagen Deposition in AlloMaxTM Acellular Dermal Matrix in Breast Reconstruction Version 8-15-12
Brief Title: Incorporation of AlloMaxTM in Breast Reconstruction Ver8-15-12
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Nevada, Las Vegas (Other)
Responsible Party: Principal Investigator, Kayvan Taghipour-Khiabani, M.D., Tenured Associate Professor, Head of Hand and Microsurgery, University of Nevada, Las Vegas
Other Study IDs: 081512
Record Dates: First submitted 2012-08-31; First posted 2012-09-05 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2015-01

CONDITIONS: Breast Cancer
Keywords: Breast reconstruction; Hydroxyproline concentration; neoangiogenesis; collagen deposition
MeSH Terms: conditions — Breast Neoplasms; Neovascularization, Pathologic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- <40 years: subjects aged less than 40 years
- 40-60 years: subjects aged 40-60years
- > 60 years: subjects aged greater than 60 years

SUMMARY:
The purpose of this study is to measure the level of AlloMax™ incorporation (cellular infiltration, collagen production, and neovascularization) in human breast reconstruction. The hypothesis is that the AlloMaxTM will have incorporation equivalent to adjacent breast capsule at the 3-4 month time point.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 - 70 yrs) who require reconstructive breast surgery with AlloMaxTM implants and agree to participate will be included in this study.

Exclusion Criteria:

* Patients who do not agree to be included in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients (18 - 70 yrs) scheduled for immediate two stage breast reconstruction with AlloMaxTM are potential subjects for this study
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2014-02; Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Hydroxyproline Concentration | 3-4 months
  Hydroxyproline will be measured in the AlloMaxTM and adjacent capsule.
Neoangiogenesis | 3-4 months
  Measure new blood vessels in AlloMaxTM and adjacent capsule
Collagen I and III | 3-4 months
  Measure collagen I and III in AlloMaxTM and adjacent capsule

CONTACTS AND LOCATIONS:
Overall Officials: Kayvan Taghipour-Khiabani, M.D., Principal Investigator — University of Nevada School of Medicine; William A Zamboni, M.D., Study Chair — University of Nevada School of Medicine
Locations (1):
- University of Nevada School of Medicine, Las Vegas, Nevada, United States